CLINICAL TRIAL: NCT00033254
Title: A Phase III Study of Conventional Radiation Therapy Plus Thalidomide (NSC#66847) Versus Conventional Radiation Therapy for Multiple Brain Metastases
Brief Title: Radiation Therapy With or Without Thalidomide in Treating Patients With Brain Metastases
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02461; RTOG-BR-0118; CDR0000069268; U10CA021661 (NIH)
Record Dates: First submitted 2002-04-09; First posted 2003-01-27 (Estimated); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Tumors Metastatic to Brain
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiotherapy; Radiation; Thalidomide

ARMS (2):
- Arm I (radiation therapy) (Active Comparator): Patients undergo radiotherapy once daily 5 days a week for 3 weeks.
  Interventions: Radiation: radiation therapy; Procedure: quality-of-life assessment
- Arm II (radiation therapy, thalidomide) (Experimental): Patients undergo radiotherapy as in arm I. Beginning on the first day of radiotherapy, patients receive oral thalidomide once daily.
  Interventions: Radiation: radiation therapy; Drug: thalidomide; Procedure: quality-of-life assessment

INTERVENTIONS:
Radiation: radiation therapy — Undergo conventional radiation therapy
  Other Names: irradiation; radiotherapy; therapy, radiation
Drug: thalidomide — Given orally
  Other Names: Kevadon; Synovir; THAL; Thalomid
  Arms: Arm II (radiation therapy, thalidomide)
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
Randomized phase III trial to compare the effectiveness of radiation therapy with or without thalidomide in treating patients who have brain metastases. Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs such as thalidomide may stop the growth of brain metastases by stopping blood flow to the tumor. It is not yet known whether radiation therapy is more effective with or without thalidomide in treating brain metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Compare the overall survival of patients with multiple brain metastases treated with radiotherapy with or without thalidomide.

II. Compare the time to tumor progression in patients treated with these regimens.

III. Compare the time to neuro-cognitive progression in patients treated with these regimens.

IV. Compare the cause of death distribution in patients treated with these regimens.

V. Compare the frequency of toxic effects of these regimens in these patients. VI. Evaluate and compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to recursive partitioning analysis class (I vs II) and planned chemotherapy after whole brain irradiation (yes vs no). Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients undergo radiotherapy once daily 5 days a week for 3 weeks. Arm II: Patients undergo radiotherapy as in arm I. Beginning on the first day of radiotherapy, patients receive oral thalidomide once daily.

Treatment with thalidomide continues for 2 years in the absence of disease progression or unacceptable toxicity. Quality of life is assessed at baseline, at completion of radiotherapy, and then every 2 months for 1 year.

Patients are followed every 2 months for 1 year, every 4 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 332 patients (166 per treatment arm) will be accrued for this study within 14.5 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed extracranial primary malignancy
* Multiple brain metastases
* At least 1 measurable brain metastasis by MRI

  * More than 4.0 cm
  * Located in midbrain or brainstem (radiosurgery ineligible)
* Performance status - Zubrod 0-1
* At least 8 weeks
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 11 g/dL*
* Hematocrit at least 35%*
* Bilirubin no greater than 1.5 mg/dL
* ALT no greater than 2 times normal
* Creatinine no greater than 1.5 mg/dL
* BUN no greater than 25 mg/dL
* No history of deep venous thrombosis
* No sensory neuropathy grade 2 or greater
* No known AIDS
* No other major medical illness or psychiatric impairments that would preclude study therapy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier method of contraception during and for at least 4 weeks after study
* No prior thalidomide
* More than 2 weeks since prior chemotherapy
* Concurrent chemotherapy allowed if more than 6 weeks past study entry (allowed during first 6 weeks of study if disease progression occurs)
* See Disease Characteristics
* No prior radiotherapy to the head or neck
* No prior radiosurgery
* Prior resection of brain metastases allowed
* No concurrent anticoagulant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2002-03; Primary Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Overall survival | Up to 6 years
  The log-rank statistic will be used.
Time to tumor progression | Date of randomization to documentation of progression, assessed up to 6 years
  Cumulative incidence model will be used to analyze the data. A multivariate Cox model analysis will be performed.
Time to neuro-cognitive progression as assessed by the Mini Mental State Exam | Up to 6 years
  Cumulative incidence model will be used to analyze the data.

SECONDARY OUTCOMES:
Cause of death distribution | Up to 6 years
Frequency of toxicities, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v3.0 | Up to 6 years
Quality of life as measured by the Spitzer Quality of Life Index (SQLI) | 6 months
Quality of life as measured by the SQLI | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Knisely, Principal Investigator — Radiation Therapy Oncology Group
Locations (1):
- Radiation Therapy Oncology Group, Philadelphia, Pennsylvania, United States